CLINICAL TRIAL: NCT01933477
Title: Strategies to Optimize Antiretroviral Therapy Services for Maternal & Child Health: the MCH-ART Study
Acronym: MCH-ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Professor Landon Myer, Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Acct#5-30539
Record Dates: First submitted 2013-08-22; First posted 2013-09-02 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: HIV
Keywords: Maternal Health; Child Health; HIV infection; Antenatal care; Postpartum care; Prevention of mother to child transmission (PMTCT); Breast feeding; Antiretrovirals
MeSH Terms: conditions — HIV Infections; Breast Feeding

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local Standard of Care (No Intervention): Arm A: Referral of post-partum women from the antenatal clinic to general adult ART services at approximately 4-8 weeks postpartum (the local current standard of care in this setting)
- MCH-focused ART services (Active Comparator): Arm B: Continued receipt of MCH-focused ART services based at the antenatal clinic throughout the period of breastfeeding. Post-partum women will only be referred to general adult ART services after the end of breastfeeding and once infants' final HIV status is determined.
  Interventions: Other: MCH-focused ART services

INTERVENTIONS:
Other: MCH-focused ART services — Post-partum women who are breast feeding will be retained in the antenatal clinic to receive continued MCH-focused ART services until after the end of breastfeeding and once infants' final HIV status is determined.
  Arms: MCH-focused ART services

SUMMARY:
The purpose of this study is to understand how to improve health care services for HIV-positive women during their pregnancy and after delivery. The study's aim is to compare two different ways of providing antiretroviral therapy for pregnant women with HIV. The study is to be conducted at the Gugulethu Midwife Obstetric Unit (MOU) in Cape Town. There are three phases of the study: Phase 1 is a cross-sectional evaluation of consecutive HIV-infected pregnant women attending their first antenatal clinic visit (n=1600); Phase 2 is an observational cohort that will follow women from Phase 1 who are eligible for ART (n=600) from the second antenatal clinic visit until the first postpartum visit; Phase 3 is a randomized trial of women from Phase 2 who are breastfeeding and will compare two different service models for delivering ART to women after they delivery their babies (n=480). For Phase 3, women who are taking ART will randomly be assigned to either (1) referral to receive ART at the nearest adult clinic at 4-8 weeks after delivery (this is currently how all women receive care in this setting) or (2) to continue to come to the antenatal clinic for ART services until the end of breastfeeding. All women will received the standard local ART services (with identical medications and medical treatment); they are different because some women will stay longer in care at the antenatal clinic. All women participating in Phase 3 will be followed through at least 2 months after they deliver.

DETAILED DESCRIPTION:
This study includes a three-phase design in which HIV-positive pregnant women are followed during the antenatal and postnatal periods. Throughout, participants will attend study measurement visits conducted separately from routine ART service appointments.

Phase 1 is a cross-sectional evaluation of consecutive HIV-infected pregnant women attending their first antenatal clinic visit seeking care at the study clinic. This phase of the study will allow characterization of the health status of the population of HIV-positive pregnant women seeking care at the Gugulethu (Midwife Obstetric Unit)MOU and the services they receive. At their first antenatal clinic visit, women will be approached to complete Informed Consent #1, including consent for abstraction of routine clinic data on obstetric and HIV-related care. As part of this cross-sectional study, participating women will complete a short questionnaire and undergo phlebotomy.

Phase 2 of the study is an observational cohort of all women who are eligible for initiation of lifelong antiretroviral therapy (following SA guidelines), from their second antenatal clinic visit until their first postpartum clinic visit (conducted within 7 days postpartum). This phase of the study will provide detailed description of ART initiation and antenatal follow-up in the population of women who will be involved in the postnatal component of the study, and be used to measure potential predictors of the primary outcome. At the second antenatal clinic visit, women from Phase 1 who are ART-eligible or who initiated ART during the pregnancy will be approached to complete Informed Consent #2, be interviewed with questionnaire on behavioral and psychosocial measures, and undergo phlebotomy. Women will complete another study measurement visit during the third trimester and again within 1 week postpartum (with study measurement visits timed to coincide with routine care appointments). At these visits, additional questionnaires and phlebotomy will be used to collect study measures.

Phase 3 of the study is a randomised trial of strategies for delivering ART to women during the postpartum period (the primary objective) with measurement of secondary outcomes during the postnatal period. Women enrolled in Phase 2 who are breastfeeding their infants will be approached to participate in the trial at the routine postpartum clinic visit (this takes place within 7 days of birth and is the only standard postpartum care for women). After completing Informed Consent #3, women will be interviewed with behavioral and psychosocial questionnaires and undergo phlebotomy for study measurements before randomization.

Randomization will be to one of two approaches to providing ART during the postpartum period to HIV-infected mothers who are breastfeeding:

* Arm A: referral to general adult ART services from approximately 4-8 weeks postpartum (the local standard of care)
* Arm B: continued receipt of ART in the antenatal clinic, as part of a MCH-focused ART service that includes primary care for HIV-exposed infants. This service only refers women to general adult ART services after the end of breastfeeding and once infants' final HIV status is determined

Women randomized to Arm A or Arm B will be asked to return for four additional study visits during the postpartum period at approximately 6 weeks, 6 months, 9 months and 12 months postpartum. Details of study measurement visits conducted in both the antenatal and postnatal periods are described below in Section 8.

For women enrolled in Phases 1 and 2 of the study, participation will not impact on any aspect of routine antenatal and obstetric care during pregnancy. Similarly, throughout the antenatal period women's HIV-related care (including PMTCT services and ART) will not be affected in any way by participation, with ART initiated according to the current standard of care. For women enrolled in Phase 3 of the study, participation will only impact on the setting and approach to providing ART services to mothers during the postpartum period, comparing immediate referral to general adult ART services versus ongoing care in MCH-focused ART services within the Gugulethu MOU.

Overall, a total of approximately 1600 HIV+ pregnant women will participate in Phase 1 of the study over 12 months. From this group, it is anticipated that approximately 400-500 HIV+ pregnant women eligible for ART will be identified as eligible for Phase 2 participation. We estimate that of the approximately 600 women on ART followed in Phase 2, approximately 480 will be eligible for and enrolled into Phase 3 and randomized to one of two postpartum ART delivery strategies.

Follow-up of all participants in Phase 3 will end at 12 months postpartum. The total length of participation will vary based on gestational age at enrollment into Phase 2, ranging from a minimum of approximately 52 weeks to a maximum of approximately 80 weeks.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* Age 18 years or older
* Documented HIV-infection according to two finger-prick rapid tests using different test types (per routine protocol in this setting) or documentation of HIV status for those women self reporting HIV diagnosis.
* Confirmed pregnancy according to urine pregnancy test, ultrasound or clinical assessment
* Able to provide informed consent for research (Informed Consent #1)

Phase 2: Subset of Phase 1 participants who are ART-eligible

* Consented and participated in Phase 1
* Documented ART eligibility based on CD4 count and/or WHO staging according to public sector testing or assessment
* Not currently using triple-drug antiretroviral therapy (women started on AZT for PMTCT during the current pregnancy are eligible) or have not used ART within the previous 6 months.
* Able to provide informed consent for research (Informed Consent #2)

Phase 3: Subset of Phase 2 participants eligible for randomization

* Consented and participated in Phase 2
* Initiated ART during the antenatal period
* Currently breastfeeding within <7 days postpartum (with an allowable window of up to 28 days postpartum)
* Willingness to be randomized and return for postnatal study visits
* Able to provide informed consent for research (Informed Consent #

Exclusion Criteria:

Individuals meeting any of the following exclusion criteria at the point in the study will be excluded:

* Not currently pregnant (Phases 1 and 2) or loss of pregnancy/neonate (Phase 3) at the time of eligibility determination
* Intention to relocate out of Cape Town permanently during the study period (Phase 2 and 3 only)
* Any medical, psychiatric or social condition which in the opinion of the investigators would affect the ability to consent and/or participate in the study (all phases), including:

  * Refusal to take ART/ARVs
  * Denial of HIV status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1554 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of (i) maternal HIV viral suppression, and (ii) maternal retention in ART services, at 12 months postpartum | Up to one year post partum follow-up for all phase 3 participants

SECONDARY OUTCOMES:
Maternal retention in care up to 12 months postpartum | Up to one year post-partum
Maternal viral suppression throughout the breastfeeding period as well as before and after cessation of breastfeeding | Up to one year post partum
Rates of HIV transmission from mother-to-child at 6 weeks and up to 12 months postpartum | Up to one year post partum
Breastfeeding practices, including duration of exclusive feeding and weaning patterns | Up to one year post partum
Acceptability of different strategies for delivering HIV care and treatment during the postpartum period | Up to one year post partum

OTHER OUTCOMES:
Subgroup analyses of the primary outcome according to participant demographic characteristics, medical history, clinical characteristics and psychosocial characteristics | up to 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Landon Myer, MBChB, PhD, Principal Investigator — University of Cape Town; Elaine J Abrams, MD, Principal Investigator — Columbia University
Locations (1):
- Gugulethu Midwife Obstetric Unit, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Weber AZ, Pellowski JA, Brittain K, Harrison A, Phillips TK, Zerbe A, Abrams EJ, Myer L. "This is My Life We are Talking About": Adaptive Strategies for HIV Care Retention and Treatment Adherence Among Postpartum Women Living with HIV in Cape Town, South Africa. Matern Child Health J. 2020 Dec;24(12):1454-1463. doi: 10.1007/s10995-020-02995-3. PMID 32816255
- [Derived] le Roux SM, Abrams EJ, Donald KA, Brittain K, Phillips TK, Zerbe A, le Roux DM, Kroon M, Myer L. Infectious morbidity of breastfed, HIV-exposed uninfected infants under conditions of universal antiretroviral therapy in South Africa: a prospective cohort study. Lancet Child Adolesc Health. 2020 Mar;4(3):220-231. doi: 10.1016/S2352-4642(19)30375-X. Epub 2020 Jan 10. PMID 31932246
- [Derived] Pellowski JA, Weber AZ, Phillips TK, Brittain K, Zerbe A, Abrams EJ, Myer L. "You must leave but I didn't want to leave": qualitative evaluation of the integration of ART into postnatal maternal and child health services in Cape Town, South Africa. AIDS Care. 2020 Apr;32(4):480-485. doi: 10.1080/09540121.2019.1659913. Epub 2019 Aug 27. PMID 31455090
- [Derived] le Roux SM, Abrams EJ, Donald KA, Brittain K, Phillips TK, Nguyen KK, Zerbe A, Kroon M, Myer L. Growth trajectories of breastfed HIV-exposed uninfected and HIV-unexposed children under conditions of universal maternal antiretroviral therapy: a prospective study. Lancet Child Adolesc Health. 2019 Apr;3(4):234-244. doi: 10.1016/S2352-4642(19)30007-0. Epub 2019 Feb 15. PMID 30773459
- [Derived] Myer L, Phillips TK, Zerbe A, Brittain K, Lesosky M, Hsiao NY, Remien RH, Mellins CA, McIntyre JA, Abrams EJ. Integration of postpartum healthcare services for HIV-infected women and their infants in South Africa: A randomised controlled trial. PLoS Med. 2018 Mar 30;15(3):e1002547. doi: 10.1371/journal.pmed.1002547. eCollection 2018 Mar. PMID 29601570
- [Derived] Sania A, Brittain K, Phillips TK, Zerbe A, Ronan A, Myer L, Abrams EJ. Effect of alcohol consumption and psychosocial stressors on preterm and small-for-gestational-age births in HIV-infected women in South Africa: a cohort study. BMJ Open. 2017 Mar 20;7(3):e014293. doi: 10.1136/bmjopen-2016-014293. PMID 28320796
- [Derived] Bernstein M, Phillips T, Zerbe A, McIntyre JA, Brittain K, Petro G, Abrams EJ, Myer L. Intimate partner violence experienced by HIV-infected pregnant women in South Africa: a cross-sectional study. BMJ Open. 2016 Aug 16;6(8):e011999. doi: 10.1136/bmjopen-2016-011999. PMID 27531735